CLINICAL TRIAL: NCT06773650
Title: Lactose Intolerance: a Guide to Proper Dietary Management, Follow-up, and Lactase Enzyme Supplementation
Brief Title: Proper Dietary Management, Follow-up, and Lactase Enzyme Supplementation for Lactose Intolerance
Status: Recruiting | Type: Observational
Sponsor: European Institute of Oncology (Other)
Responsible Party: Sponsor
Other Study IDs: UID 4675
Record Dates: First submitted 2025-01-09; First posted 2025-01-14 (Actual); Last update posted 2025-01-14 (Actual); Status verified 2025-01

CONDITIONS: Lactose Intolerant; Lactose Malabsorption; Lactose Intolerance
MeSH Terms: conditions — Lactose Intolerance

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Patients completing online survey: The online survey aims to reach a representative sample of the Italian population to identify their knowledge regarding Lactose Intolerance
  Interventions: Other: Completion of online survey

INTERVENTIONS:
Other: Completion of online survey — The online survey aims to reach a representative sample of the Italian population to identify their knowledge regarding LI

SUMMARY:
Lactose intolerance (LI) is considered the clinical syndrome caused by lactose malabsorption (LM).

It is possible to identify four causes of lactase deficiency defining four different types of LM: primary (genetic), secondary (acquired), congenital (alactasia), and developmental (in premature infants, so reversible).

The aim of this protocol is to investigate through an anonymous online survey the knowledge of the Italian population on clinical, pathophysiological, diagnostic and therapeutic issues of lactose intolerance. Data collected will be divulgated through a publication for both people with IL and nutritionists, enriched with tables and flow charts, to improve the knowledge on lactose intolerance and to support people suffering from this condition. The results of this survey will guide subjects suspected of suffering from lactose intolerance towards a correct diagnosis and a better management.

ELIGIBILITY:
Inclusion Criteria:

* Subjects must be adults (≥18 years of age)
* Willingness to complete the online survey

Exclusion Criteria:

* Subjects <18 years of age
* Subjects not available to answer the online survey

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The online survey aims to reach a representative sample of the Italian population to identify their knowledge regarding Lactose Intolerance
Sampling Method: Probability Sample
Enrollment: 385 (Estimated)
Dates: Start 2025-01-08 (Actual); Primary Completion 2026-01 (Estimated); Study Completion 2026-01 (Estimated)

PRIMARY OUTCOMES:
Evaluation of knowledge of the Italian population on lactose intolerance | 3 months
  The aim of this protocol is to investigate through an anonymous online survey the knowledge of the Italian population on clinical, pathophysiological, diagnostic and therapeutic issues of lactose intolerance

CONTACTS AND LOCATIONS:
Locations (1):
- European Institute of Oncology, Milan, Italy

IPD SHARING:
Plan to Share IPD: No